CLINICAL TRIAL: NCT05776082
Title: Association of Cardiovascular Health During Pregnancy With Perinatal Outcomes---a Birth Cohort Study
Brief Title: Association of Gestational Cardiovascular Health With Pregnancy Outcomes
Status: Recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20230053-R
Record Dates: First submitted 2023-02-23; First posted 2023-03-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-04

CONDITIONS: Pregnant Women
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, saliva, placenta and umbilical cord blood from pregnant women will be collected for testing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire survey and specimen collection — Questionnaire survey, clinical follow-up and specimens collection.

SUMMARY:
Pregnancy is a critical period for cardiovascular health risk assessment and interventions to reduce the incidence of cardiovascular disease in both mother and child generations. Recently, the American Heart Association proposed the latest cardiovascular health assessment indicator "Life's Essential 8". However, there is still a lack of application data for pregnant women. This project intends to explore the application potential of Life's Essential 8 in cardiovascular health assessment of pregnant women and establish appropriate gestaional cardiovascular health standards.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age: 20-49 years;
* Natural conception;
* Single pregnancy;
* Plan to have routine prenatal examinations and give birth in the research center;

Exclusion Criteria:

* Have diseases that affect metabolic function or even threaten the life of the mother and fetus before pregnancy;
* Assisted reproduction;
* Multiple pregnancy;
* Fetus has a known deformity or genetic defects;
* Incomplete clinical data.

Ages: 20 Years to 49 Years | Sex: Female
Age Groups: Adult
Study Population: This project intends to recruit pregnant women who go to the research center for routine prenatal examination and give birth.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal outcomes | Through delivery completion, up to 42 weeks
  Including pregnancy-induced hypertension, preterm delivery, abortion, delivery way and so on. They are diagnosed by clinicians and the data is gathered from medical records.
Neonatal outcomes | Through delivery completion, up to 42 weeks
  Birth weight（in gram), birth height (in centimetre), gestational week (in week) and other neonatal diseases. They are diagnosed by clinicians and the data is gathered from medical records.

CONTACTS AND LOCATIONS:
Locations (3):
- China (2):
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang
- Rwanda Society of Obstetricians and Gynecologists, Kigali, Rwanda